CLINICAL TRIAL: NCT01970800
Title: The Role of Igf-1 Generation Test in Diagnosis and Treatment of Short Stature
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Nature of study was changed from ACT to retrospective chart review
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10/01/VA03
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Short Stature
Keywords: IGF-1; Short Stature; GH
MeSH Terms: conditions — Dwarfism | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: This study was changed to a retrospective chart review. There was no prospective component.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Growth hormone, injections (Experimental): Growth hormone injection 0.3mg/kg/week dailY
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — Will obtain daily injections and will evaluate the IGF-1 and IGFBP3 every 3 months
  Other Names: Nutropin AQ

SUMMARY:
The purpose of the study is to evaluate the predictive value of IGF-1 generation test for growth velocity during GH treatment for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide written informed consent
* Prepubertal males and females form 5- 11years old
* Bone age <11 years in males and <9 years in females
* Height SD score<-2.25SD in males and females
* IGF-1SD score <-1SD in both males and females
* Peak GH level after stimulation >10ng/ml

Exclusion Criteria:

* History of prior chemotherapy and or radiation
* Active neoplasm
* Pediatric patients with closed epiphyses
* Prader-Willi syndrome, Turner syndrome or any other genetic or chromosomal anomaly
* Treatment with inhaled or systemic steroids
* BMI <5th percentile or >95th percentile
* Tanner 2 at clinical or biochemical examination by ultrasensitive LH and FSH

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Outcome measurement | one year
  Growth velocity after treatment with appropriate growth hormone doses

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Ten, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States